CLINICAL TRIAL: NCT06568380
Title: Investigation of Norovirus Infection Incidence According to the Presence of Fecal Bacteriophages After Oyster Consumption : Randomized Controlled Clinical Trial - VIROYSTER
Brief Title: Validation of a Boindicator as Monitoring Tool for Oyster Norovirus Outbreak
Acronym: VIROYSTER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study abandoned before authorization obtained
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2019-A01763-54
Record Dates: First submitted 2019-09-23; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Gastroenteritis Norovirus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Noro+ Phage+ (Experimental): Oysters positives for both norovirus genome and infectious bacteriophages
  Interventions: Other: Oyster consumption
- Noro+ Phage- (Experimental): Oysters positives for norovirus genome and negatives for infectious bacteriophages
  Interventions: Other: Oyster consumption
- Noro- Phage+ (Experimental): Oysters negatives for norovirus genome and positives for infectious bacteriophages
  Interventions: Other: Oyster consumption
- Noro- Phage- (Placebo Comparator): Oysters negatives for both norovirus genome and infectious bacteriophages
  Interventions: Other: Oyster consumption

INTERVENTIONS:
Other: Oyster consumption — Volunteers consume one of the four panel of oysters (Noro+Phage+, Noro+Phage-, Noro-Phage+ and Noro-Phage-).

SUMMARY:
Noroviruses are responsible for 700M of annual cases of gastroenteritis, of which 15M are directly related to the consumption of contaminated food, including oysters. Current regulations do not require control of human noroviruses in shellfish. However, an ISO standard recommended to detect their genome in high-risk foodstuffs. However, presence of viral genome doesn't testify to the presence of infectious particles. Routine application of this standard would therefore wrongly lead to the withdrawal of shellfish from market, since norovirus genomes are widely found in the environment and in food without indicating a viral risk. Given the difficulty of cultivating human noroviruses in vitro and thus of discriminating infectious particles from non-infectious particles only based on genome detection, it is necessary to identify an indicator of the infectious nature of these pathogenic viruses. To be suitable, the indicator must first be associated with the presence of norovirus genome in the environment. This is the case of fecal bacteriophage F-specific RNA. Since bacteriophages are cultivable in the laboratory, it is easy to estimate the proportion of genomes of these bacteriophages corresponding to infectious particles. To confirm this indicator, it is necessary to demonstrate a relationship between the presence of infectious bacteriophages with that of infectious norovirus. This is only estimable by the occurrence of a gastroenteritis after consumption of a contaminated food by humans. We propose this randomized controlled clinical trial to evaluate the incidence of norovirus infection after consumption of oysters free from or containing infectious F-specific RNA bacteriophages.

The purpose of this study is to evaluate if norovirus infections incidence is significantly weak after the consumption of oysters free of F-specific infectious RNA bacteriophages, compared to the consumption of oysters containing these same infectious bacteriophages.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Health status
* No seafood allergy
* Nancy city residents

Exclusion Criteria:

* Recent gastroenteritis (<6 months)
* Fragile health person proximity
* Oysters consumption during the study
* Pregnancy or breastfeeding
* "nonsecretor" phenotype

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Norovirus concentration in feces (genome copy number/grammes of feces) | Baseline (J0) and during symptoms if any or within 36-60 hours after consumption in another case
  A norovirus genome augmentation may indicate virus replication
Gastroenteritis symptoms | within 3 days after consumption
Immunoglobulin A (IgA) detection in feces | within 3-5 days after consumption
  In case of asymptomatic infection, IgA are secreted

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Gantzer, Pr, Study Director — LCPME -UMR Université de Lorraine/CNRS
Locations (1):
- CHRU Nancy, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided